CLINICAL TRIAL: NCT07347145
Title: Clinical Evaluation of Hair Loss and Hair Growth Human Volunteers Following a Double-blind, Placebo-controlled, 2:1 Randomized Trial of 'Olistic Next Women'
Brief Title: Clinical Evaluation of a Nutraceutical Supplement for Hair Growth, Hair Loss and Skin Improvement in Human Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olistic Research Labs S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-ON-02
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Early Female Pattern Hair Loss (FPHL)
MeSH Terms: interventions — Minerals; Plant Extracts; Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olistic Next Women (Active Comparator)
  Interventions: Dietary Supplement: Drinkable multifactorial food supplement containing vitamins, minerals, plant extracts, amino acids, and other bioactive compounds, formulated to support hair growth and scalp health in women.
- Placebo Arm (Placebo Comparator)
  Interventions: Other: Placebo control

INTERVENTIONS:
Dietary Supplement: Drinkable multifactorial food supplement containing vitamins, minerals, plant extracts, amino acids, and other bioactive compounds, formulated to support hair growth and scalp health in women. — Drinkable multifactorial food supplement in liquid form, administered once daily in a 25 mL single-dose vial, for a duration of 180 days. The formulation contains a combination of vitamins, minerals, plant extracts, amino acids, and other bioactive compounds designed to support hair growth and scalp health in women.
  Arms: Olistic Next Women
Other: Placebo control — Drinkable formulation consisting of an excipient formulation designed to mimic the organoleptic properties of the active product, reproducing its color and texture while achieving a highly similar taste profile.
  Arms: Placebo Arm

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Olistic Next Women, a nutraceutical supplement, in women experiencing beginning of female pattern hair loss (FPHL).This 6-month, double-blind, placebo-controlled, 2:1 randomized clinical trial investigates whether daily supplementation with Olistic Next Women leads to significant improvements in hair parameters compared to placebo. The study also monitors the tolerability and safety of the product throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with female pattern hair loss
* 45-65 years
* Signed informed consent
* The study participant is in good general condition for her age and does not currently have any active diseases that, in the opinion of the investigator, justify exclusion from the study.

Exclusion Criteria:

* Known or documented intolerance/allergy to any of the ingredients of the study product
* Chronic wounds, erosions, pre-existing infected skin or inflammation in the study area
* Suspected non-compliance
* Late onset acne
* Hirsutism
* Any systemic immunosuppressant given within the 12 months prior to the study (e.g. systemic Prednisolone in high doses, Azathioprine, Metothrexate etc.)
* Locally (in the study area) applied products/medicaments which in the opinion of the investigator could lead to an influence of the study results (e.g. topical minoxidil, caffeine etc.)
* Systemically administered products and medicaments which in the opinion of the investigator could lead to an influence of the study results (e.g. hormone-influencing medicaments, medicaments which frequently lead to hypertrichosis or hair loss etc.)
* Subjects receiving stable hormone replacement therapy (HRT) for <6 months prior to screening will be excluded.
* Subjects who follow an exclusively or mainly vegan diet
* Known or documented Gluten intolerance
* Lactose intolerance
* Hyperthyroidism
* Subjects with hypothyroidism with non-stable thyroid-stimulating hormone (TSH) levels will be excluded.
* Other diseases of the scalp which in the opinion of the investigator could lead to an influence of the study results (e.g. Lichen planus, Psoriasis capitis, scarring alopecia etc.)
* Participation in a clinical trial/study
* Participation in a clinical trial/study within the last 30 days
* Deviations from the norm in the following laboratory values in the blood test of the screening visit: zinc, ferritin, selenium, folic acid, vitamin B12, TSH, and CRP. (Only at Baseline)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Increase in hair density | From enrollment to the end of treatment at 180 days.
  From phototrichogram on the Sagittal midline area of the scalp.

SECONDARY OUTCOMES:
Change in hair shedding | From enrollment to the end of treatment at 180 days.
  Hair shedding will be assessed by collecting shed hairs during a standardized washing and combing procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- CentroDerm, Wuppertal, Barmen, Germany

IPD SHARING:
Plan to Share IPD: No